CLINICAL TRIAL: NCT05763745
Title: Bedside Ultrasonic Assessment for Gastric Content in Patients With Upper GI Bleeding
Brief Title: Bedside Ultrasonic Assessment for Gastric Content in Patients With Upper GI Bleeding Undergoing Endoscopy
Status: Completed | Type: Observational
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Other Study IDs: 5220358
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Upper GI Bleeding; Point of Care Ultrasound; Upper Endoscopy; Gastric Content; GI Bleed
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Point of Care Ultrasound
  Interventions: Diagnostic Test: Point of Care Ultrasound

INTERVENTIONS:
Diagnostic Test: Point of Care Ultrasound — Use Point of Care Ultrasound to evaluate the gastric content/bleed prior to upper endoscopy

SUMMARY:
Emerging studies have evaluated POCUS (Point of Care Ultrasound) for assessing of gastric content prior to anesthesia to reduce the risk of aspiration and demonstrated that POCUS can accurately identify presence of gastric food or fluid. Despite accumulating studies evaluating POCUS as a diagnostic modality to evaluate for gastric food content prior to anesthesia, there is no study to date that has evaluated the role of POCUS prior to endoscopy among patients with upper GI bleeding. Therefore, this study is to evaluate the diagnostic accuracy of POCUS for retained gastric content prior to endoscopy among patient hospitalized/admitted with upper GI bleeding. This study would take place at Loma Linda University Medical Center. Subjects will be any one who has upper GI bleed required EGD and age of greater than 18 years old. The study will plan for 1 year or reach 50 patients (whichever one comes first). In addition, subjects will be recruited from ED, ICU, Medicine ward by the PI, SubPI, and Collaborators. Subject will received ultrasound up to 6 hours prior the start of endoscopy. The location of Ultrasound would either take place at GI lab prior to scope or at the ward prior to transportation to GI lab or at ICU prior to endoscopy. The ultrasound would focus upper abdomen area and look for antrum. the result will be immediately read before endoscopy and fill out on the sheet before the endoscopy. Patient then proceed with endoscopy. At the end of the scope, the researcher will ask the endoscopist questions regarding how well they could see each part of the stomach in order to complete the study. Both results are compared between US and Endoscopy. Endoscopist is blinded in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18
2. patient presents with hematemesis
3. and/or melena
4. and/or hematochezia accompanied by hemodynamic changes (pulse >100/min and/or systolic blood pressure <100/min)
5. Patient is scheduled for upper endoscopy due to the above.

Exclusion Criteria:

1. Decline consent for study
2. Patients with last solid meal <6 hours and clear liquids <2 hours prior to the endoscopy
3. Prior surgery in the stomach
4. Patient has duodenum, Ileus, or bowel obstruction
5. patient has history of gastric cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age >18 admitted with upper GI bleeding defined by symptoms of hematemesis, melena, and/or hematochezia accompanied by hemodynamic changes (pulse >100/min and/or systolic blood pressure <100/min) scheduled for upper endoscopy.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
measurement is gastric food content/blood. | after obtaining informed consent and prior to endoscopy being conducted.
  Ultrasound would be conducted on upper abdomen to evaluate the presence of blood and/or food in the stomach. The result would divided into empty (no food), small and large. ultrasound mainly evaluate the antrum area to see whether it is dilated/distended or not. if it is collapsed, then it is considered empty. If it is largely dilated, it would be considered large.

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: Undecided